CLINICAL TRIAL: NCT03889353
Title: Is Mental Motor Imagery Training Using "GHOST", a Novel BCI-VR Feedback System (Brain Computer Interface and Virtual Reality) Efficient and Safe for Pain Relief in Phantom Limb Pain After Upper Limb Amputation or Brachial Plexus Lesion
Brief Title: Brain Computer Interface and Virtual Reality (BCI-VR) for Pain Treatment
Acronym: GHOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC17_0417
Record Dates: First submitted 2019-03-08; First posted 2019-03-26 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCI sessions (Experimental): up to 3 test sessions (Day-30) to eliminate BCI illiteracy, then 10 rehabilitation sessions of 90 minutes (Day 1-Day 5 and Day 8-Day 12) - Session content : Guided training - Control of an avatar (VR, first person view) of the affected limb by motor mental imagery decoded by a brain computer interface.
  Interventions: Device: BCI sessions

INTERVENTIONS:
Device: BCI sessions — up to 3 test sessions (D-30) to eliminate BCI illiteracy, then 10 rehabilitation sessions of 90 minutes (D1-D5 and D8-D12) - Session content : Guided training - Control of an avatar (VR, first person view) of the affected limb by motor mental imagery decoded by a brain computer interface.

SUMMARY:
Pilot Interventional study with minimal risks and constraints, prospective, monocentric. Safety and Efficacity evaluation of a Novel Medical Device.

DETAILED DESCRIPTION:
Upper limb's phantom pain, due to amputation or to injury of the brachial plexus are possibly due to maladaptive CNS (central nervous system facility) plasticity and thus could be decreased by retraining the sensorimotor cortex using Mental Motor Imaging guided through a novel BCI-RV feedback system : "Ghost". The aim of this study is to evaluate safety and efficacy of this BCI pain treatment developed by our team.

ELIGIBILITY:
Inclusion Criteria:

* Neuropathic pain / Phantom limb pain
* Mean pain score >3 centimeter
* Permanent pain
* If Plexus Brachial injury : > 6 month
* If Amputation : at least at wrist level
* Motor and Sensory deficit : complete or incomplete
* Informed consent
* Public Health Insurance

Exclusion Criteria:

* MRI contraindication
* Subject included in another interventional study
* Pregnant women
* Majors under guardianship or curatorship or safeguard of justice
* History of associated head injury or any other neurological pathology altering the sensorimotor cerebral system or cognitive abilities and higher functions.
* Presence of other lesions of the peripheral nervous system that may induce associated neuropathic pain.
* Head trauma associated altering somatosensory system or cognitive abilities and higher functions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of BCI intervention on mean daily pain | month 6
  Determination by curve fitting technique (regression analysis) of the peak effect and calculation of the rate of improvement: success if> 30%

SECONDARY OUTCOMES:
Evaluate the effectiveness of the BCI intervention on paroxysmal pains | 60 days from day -30 to day + 30 , once a week from Month 1 to month 6
  duration of the paroxysmal pains
Evaluate the effectiveness of the BCI intervention on paroxysmal pains | 60 days from day -30 to day + 30 , once a week from Month 1 to month 6
  the intensity of paroxysmal pains This scale measures the intensity of paroxysmal pain. It is a self-assessment. Scores measured with Visual Analog Score.
  The scale is graded from 0 (no pain) to 10 (most intense pain the patient can imagine).
  The value 10 (maximum) is the worst result. There is no combination of sub-ranges to compute the score
Evaluate the effectiveness of the BCI intervention on paroxysmal pains | 60 days from day -30 to day + 30 , once a week from Month 1 to month 6
  the frequency of paroxysmal pains
Evaluate the effect of the intervention on quality of life: SF36 | Day 1, 12, 90, 180
  SF36 Questionnaire quality of life For each question, an algorithm allows the calculation of scores to obtain a number between 0 (zero quality - worse outcome) and 100 (maximum quality).
Evaluate the effect of the intervention on anxiety and depression | Day 1, 12, 90, 180
  HAD questionnaire : Hospital Anxiety and Depression scale It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), resulting in two scores (maximum score of each score = 21).
  To detect anxious and depressive symptoms, the following interpretation can be proposed for each of the scores (A and D):
  * 7 or less: lack of symptomatology
  * 8 to 10: doubtful symptomatology - 11 and more: definite symptomatology.
evaluating cortical plasticity | Day 1, 12, 30
  MRI analysis the physiopathological mechanisms governing phantom pain
evaluating cortical plasticity | Day 1, 12, 30
  EEG analysis the physiopathological mechanisms governing phantom pain
Evaluate the performance of subjects to control the neurofeedback system | Day 1, 12, 30
  Motor Imagery Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes Uh, Nantes, France

IPD SHARING:
Plan to Share IPD: No